CLINICAL TRIAL: NCT03908398
Title: Comparison Process-oriented and Outcome-oriented Visual Assessments for the Evaluation of Hospital Cleanliness
Brief Title: Process-oriented and Outcome-oriented Visual Assessments
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CW18285B
Record Dates: First submitted 2019-04-03; First posted 2019-04-09 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Hospital Cleanliness
Keywords: ATP bioluminescence; Visual assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to compare the effectiveness of outcome-oriented visual assessment and process-oriented visual assessment using ATP bioluminescence test as a comparator in order to find out which method can be used to assess hospital cleanliness.

DETAILED DESCRIPTION:
This study was conducted in a 17-bed adult medical intensive care unit at a medical center during December 2019 to December 2020. First of all, high-touch room surfaces were selected in patient rooms, including bed rails / controls, light switch, IV pump control, feeding pump control, monitor control, bedside table handle, call button, IV pole (grab area) and suction machine control. Then, Areas to be sampled on those high-touch room surfaces were identified. Whenever the housekeepers started to do terminal cleaning after patients were transferred or discharged, the researcher also started to observe directly the practices of cleaning at the same time and recorded "cleaned" if surfaces were cleaned and disinfected properly. Then, the researcher inspected surfaces and recorded "clean" if surfaces were free of dust, debris, and stains immediately after terminal cleaning.Ten minutes after terminal cleaning, Hygiena Ultrasnap Surface ATP test was performed to swab a standard area of 10 square centimeters on specific surfaces. After completing sampling, swabs were replace back in swab tube and all liquid in bulbs was expelled to activate the reaction. Once activated, samples were read right after shaking swab tube for 5-10 seconds.

ELIGIBILITY:
Inclusion Criteria:

* the environmental surfaces immediately after patients are discharged

Exclusion Criteria:

* no

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: We compare the degrees of agreement between the ATP data, process-oriented visual assessment scores and outcome-oriented visual assessment scores after environmental cleaning.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
ATP DATA | 10 minutes after environmental cleaning
  ATP bioluminescence test
score of process-oriented visual assessments | immediately after environmental cleaning
  There are ten environment surfaces. Whenever the housekeepers start to do terminal cleaning after patients are transferred or discharged, the researcher also start to observe the practices of cleaning at the same time and score "one point" if one surface is cleaned and disinfected properly. The total of the score is ten.
score of outcome-oriented visual assessments | immediately after environmental cleaning
  There are ten environment surfaces. Whenever the housekeepers start to do terminal cleaning after patients are transferred or discharged, the researcher also start to observe directly the cleanliness of the environment surfaces at the same time and score "one point" if one surface is clean visually. The total of the score is ten.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chun Chen, MS, Study Chair — Taichung Veterans General Hospital Infection Control Center
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No